CLINICAL TRIAL: NCT05896293
Title: Kisspeptin Administration Subcutaneously to Patients With Reproductive Disorders
Brief Title: Kisspeptin Administration Subcutaneously to Patients With IHH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephanie B. Seminara, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FD007843
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: Hypogonadotropic Hypogonadism; Kisspeptin; Idiopathic Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism; Idiopathic Hypogonadotropic Hypogonadism | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- kisspeptin pump (Experimental): SC administration of kisspeptin for two weeks (pulsatile, every 60-240 minutes); administration of a single shot of leuprolide acetate (previously GnRH was used in this study)
  Interventions: Drug: kisspeptin 112-121; Drug: leuprolide acetate

INTERVENTIONS:
Drug: kisspeptin 112-121 — SC administration of kisspeptin for two weeks (pulsatile, every 60-240 minutes)
  Other Names: metastin 45-54
Drug: leuprolide acetate — Single SC bolus

SUMMARY:
The goal of this study is to see whether kisspeptin, a naturally occurring hormone, can stimulate the release of other reproductive hormones in men and women with idiopathic hypogonadotropic hypogonadism (IHH). The investigators are also examining whether kisspeptin can help women release eggs from their ovaries. Kisspeptin will be administered SC for two weeks in a pulsatile fashion. Ultrasound monitoring of ovarian follicular growth (for women) and frequent blood sampling (every 10 minutes for up to 70 minutes) will be performed to assess the physiologic response to kisspeptin over time.

Funding Source: FDA OOPD

DETAILED DESCRIPTION:
Assignment: All study subjects will undergo the same interventions.

Delivery of Interventions:

* Each subject will undergo a review of their medical history, physical exam, and screening laboratories.
* A single SC injection of leuprolide acetate may be administered approximately six days before kisspeptin administration. (Previously administration of Gonadotropin Releasing Hormone (GnRH) was used in this study.)
* A pelvic ultrasound will be performed on women to assess baseline follicular size.
* A pump will be placed to administer pulsatile SC kisspeptin for two weeks.
* During the course of kisspeptin administration, subjects will

  * Undergo q10 min blood sampling (approximately 10 sessions, 70 minutes each)
  * For women, undergo pelvic ultrasounds (approximately 4 sessions)
* Optional q10 min sampling up to 8 hours may take place before and after the course of kisspeptin

ELIGIBILITY:
Inclusion Criteria:

* Congenital IHH

  o Confirmed diagnosis by medical provider supported by low sex steroids in the setting of low or inappropriately normal gonadotropins
* Normal blood pressure (systolic BP < 140 mm Hg, diastolic < 90 mm Hg)
* No current or recent use of a medication that, in the opinion of a study investigator, can modulate the reproductive axis or willing to complete an appropriate washout for that particular medication and method of administration

Exclusion Criteria:

* Any condition (medical, mental, or behavioral) that, in the opinion of a study investigator, would likely interfere with participation in/completion of the protocol
* Excessive alcohol consumption (>10 drinks/week) and/or active use of illicit drugs

  o Any active use of marijuana will be evaluated by a study medical professional to determine if it may impact study participation.
* Pregnant or trying to become pregnant
* Breast feeding
* History of: bilateral oophorectomy (both ovaries were removed), breast cancer, thromboembolic disease, coronary artery disease, stroke, thrombophilic disorders, or undiagnosed abnormal genital bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Average change in luteinizing hormone (LH) pulse amplitude | 2 weeks
  Average difference in LH amplitude after the first dose of kisspeptin (day 1) compared to the last dose of kisspeptin (day 15)

SECONDARY OUTCOMES:
Percentage of female participants who demonstrate achievement of a mature follicle or show evidence of ovulation | 2 weeks
  Percentage of female participants that develop a mature follicle or ovulate. Mature follicle achievement is defined as evidence of a follicle with maximum diameter ≥18 mm. Evidence of ovulation is defined as detection of a corpus luteum on ultrasound in combination with elevated progesterone level.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No